CLINICAL TRIAL: NCT04133272
Title: Registry of Ehlers-Danlos Syndrome That Collects Clinical, Functional, Genetic, Genealogical, Imaging, Surgical, Treatment, Quality of Life Data. Data Are Linked to Patients' Biological Samples, When Available
Brief Title: Registry of Ehlers-Danlos Syndrome
Acronym: RED
Status: Recruiting | Type: Observational
Sponsor: Luca Sangiorgi (Other)
Responsible Party: Sponsor-Investigator, Luca Sangiorgi, Head of Department of Rare Skeletal Disorders, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: 21611/2014
Record Dates: First submitted 2019-10-14; First posted 2019-10-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ehlers-Danlos Syndrome
Keywords: Disease Registry; Natural History Study; Disease Evolution; Genotype-Phenotype Correlation
MeSH Terms: conditions — Ehlers-Danlos Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — Whole peripheral blood, DNA, lymphocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ehlers-Danlos Syndrome patients: The group comprises all patients affected by Ehlers-Danlos Syndrome, including prenatal and fetal diagnosis of Ehlers-Danlos Syndrome

SUMMARY:
RED is a retrospective and prospective registry, finalized for care and research purposes. It is articulated in main sections - strongly related and mutually dependent on each other - corresponding to different data domains: personal information, clinical data, genetic data, genealogical data, surgeries, etc.

This approach has been developed to corroborate and integrate data from different sources and evaluating several aspects of diseases and to correlate genetic background and phenotypic outcomes, in order to better investigate disease pathophysiology. Due to legal requirements, institutional directives and organizational issues, we are unable to include individuals residing outside Italy in the registry at this time. We are currently engaged in the preparation of a recruitment process for individuals residing outside Italy.

DETAILED DESCRIPTION:
The traditional method of collecting patient information is often chaotic, inconvenient and sometimes even unsafe, particularly when dealing with rare diseases. In 2014, the need to simplify the diagnostic process and to overcome the difficulties of data storage and analysis, led to the suggestion of implementing the Registry of Ehlers-Danlos Syndrome (RED).

The RED relies on an IT platform named Genotype-phenotype Data Integration platform - GeDI. This solution was developed through a collaboration between Rare Skeletal Disease Department and a local software company (Dilaxia) and is General Data Protection Regulation (GDPR)-compliant, multi-client and web-accessible. It has been designed according to current medical informatics standards, including the Orphanet code, the International Classification of Diseases (ICD), the Human Genome Variants Society, aiming to follow FAIR (Findability Accessibility Interoperability Reusability) principles. GeDI is continuously being implemented to improve the management of people with Ehlers-Danlos Syndrome and to assist researchers in analysing the information collected. RED is divided into the following main sections:

* Personal data: it comprises general information, birth details and residence data;
* Patient data: including the patients internal code, the hospital code and other patient details;
* Diagnostic Process: the diagnosis, the status (affected, suspected, etc.), age at diagnosis, comorbidities, allergies, etc.;
* Genogram: a tool for designing the family transmission of the disease, alongside information on the disease status of all relatives included;
* Clinical events: it records a long list of signs and symptoms of Ehlers-Danlos Syndrome as well as several additional items to describe the disease
* Genetic Analysis and Alteration: including analytical technique, sample information, analysis duration, etc. This section also comprises detailed information on any detected pathological variants (e.g. gene, international reference, DNA change, protein change, genomic position, etc.);
* Visits: this section includes visit type (genetic, orthopedic, rehabilitation, pediatric, etc.), the date of the visit, prescriptions, imaging, etc.;
* Treatments: this section comprises information of a wide range of treatments including pharmacological, devices, supplements, and other treatments such as psychological, nutritional, etc.;
* Surgeries: this section contains information on the type of surgeries, the age of the patients, the site/localization of the procedures, etc.
* Documents: this repository allow us to store all types of documents (radiological reports, imaging, consents, clinical reports, etc.);
* Consents: this section provides a comprehensive overview of all consents collected, including the collection date;
* Samples: this section includes information on the samples, like the type, date of collection, etc.
* PROs: this section collects information on patients reported outcomes such as the quality of life or ABC scale.

ELIGIBILITY:
Inclusion Criteria:

* All Ehlers-Danlos Syndrome patients, including prenatal and fetal diagnosis of Ehlers-Danlos Syndrome

Exclusion Criteria:

* Any condition unrelated to Ehlers-Danlos Syndrome

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by Ehlers-Danlos Syndrome. The Registry will include also data on fetuses (prenatal and abortion)
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Natural History and Epidemiology in terms of clinical, genetic and functional evaluation | 25 years
  To maintain an established registry in order to assess epidemiology and natural history.
  Collection of:
  1. physical examinations data: assessment of type of the disease (according to Orphanet types)
  2. orthopedic and functional data: stature (cm), weight (kg), Beighton score, pain score (numeric scale), presence cardiac lesion (ultrasound)
  3. surgical procedures: type, number and site of surgeries disease-related and age at surgeries
  4. genetics background: target gene, type of mutation, type of variant detected, clinical significance
  5. family history: inheritance in maternal or paternal line
  6. treatment information: pharmacological, devices, supplements, and other treatments
  Clinical, orthopedic, surgical, treatment and functional features are updated at each follow up. Clinical reports, medical charts, genetic report and imaging are the primary sources of data.

SECONDARY OUTCOMES:
Genotype-Phenotype Correlation among clinical features and molecular background | 25 years
  The secondary outcome comprises the correlation between genotype and phenotype. This includes but is not limited to clinical features and genetic background. This will be pursued using the information collected during visits and follow-ups and the genetic information resulting from molecular investigations

OTHER OUTCOMES:
Longitudinal study of disease (including prospective and retrospective data) | 25 years
  This outcome aims to investigate the Ehlers-Danlos Syndrome trend during time. This will be evaluated within the families and among the families.
  Main clinical features, such as height (cm), pain (numeric scale) and other variables will be collected both retrospectively and prospectively. An evaluation of these parameters will be performed at each visit to keep track on the progression of clinical manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Sangiorgi, MD, PhD, MS, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Ritelli M, Rovati C, Venturini M, Chiarelli N, Cinquina V, Castori M, Colombi M. Application of the 2017 criteria for vascular Ehlers-Danlos syndrome in 50 patients ascertained according to the Villefranche nosology. Clin Genet. 2020 Feb;97(2):287-295. doi: 10.1111/cge.13653. Epub 2019 Nov 3. PMID 31600821
- [Background] Ghali N, Sobey G, Burrows N. Ehlers-Danlos syndromes. BMJ. 2019 Sep 18;366:l4966. doi: 10.1136/bmj.l4966. No abstract available. PMID 31533917
- [Background] Black CM, Gathercole LJ, Bailey AJ, Beighton P. The Ehlers-Danlos syndrome: an analysis of the structure of the collagen fibres of the skin. Br J Dermatol. 1980 Jan;102(1):85-96. doi: 10.1111/j.1365-2133.1980.tb05675.x. PMID 7378285
- [Background] Beighton P. Ehlers-Danlos syndrome. Ann Rheum Dis. 1970 May;29(3):332-3. doi: 10.1136/ard.29.3.332. No abstract available. PMID 5432600
- [Background] Benistan K, Gillas F. Pain in Ehlers-Danlos syndromes. Joint Bone Spine. 2020 May;87(3):199-201. doi: 10.1016/j.jbspin.2019.09.011. Epub 2019 Sep 25. No abstract available. PMID 31562935
- [Background] Hausser I. Diagnosis of Ehlers-Danlos syndrome: data deficiency still does not allow establishment of a complete history of the disease and its pathomechanisms. Br J Dermatol. 2020 Mar;182(3):535-536. doi: 10.1111/bjd.18373. Epub 2019 Aug 20. No abstract available. PMID 31432500
- [Background] Jesudas R, Chaudhury A, Laukaitis CM. An update on the new classification of Ehlers-Danlos syndrome and review of the causes of bleeding in this population. Haemophilia. 2019 Jul;25(4):558-566. doi: 10.1111/hae.13800. Epub 2019 Jun 10. PMID 31329366
- [Background] De Baets S, Calders P, Verhoost L, Coussens M, Dewandele I, Malfait F, Vanderstraeten G, Van Hove G, Van de Velde D. Patient perspectives on employment participation in the "hypermobile Ehlers-Danlos syndrome". Disabil Rehabil. 2021 Mar;43(5):668-677. doi: 10.1080/09638288.2019.1636316. Epub 2019 Jul 9. PMID 31287330
- [Background] Copetti M, Morlino S, Colombi M, Grammatico P, Fontana A, Castori M. Severity classes in adults with hypermobile Ehlers-Danlos syndrome/hypermobility spectrum disorders: a pilot study of 105 Italian patients. Rheumatology (Oxford). 2019 Oct 1;58(10):1722-1730. doi: 10.1093/rheumatology/kez029. PMID 30783660
- [Background] Mu W, Muriello M, Clemens JL, Wang Y, Smith CH, Tran PT, Rowe PC, Francomano CA, Kline AD, Bodurtha J. Factors affecting quality of life in children and adolescents with hypermobile Ehlers-Danlos syndrome/hypermobility spectrum disorders. Am J Med Genet A. 2019 Apr;179(4):561-569. doi: 10.1002/ajmg.a.61055. Epub 2019 Jan 31. PMID 30703284
- See also: Institutional webpage of Registries For Rare Hereditary Diseases — https://www.ior.it/en/curarsi-al-rizzoli/registries-rare-hereditary-diseases